CLINICAL TRIAL: NCT04446000
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous CSL730 in Healthy Adult Subjects
Brief Title: Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneous CSL730 in Healthy Adult Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of clinical viability
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSL730_1002; 2019-001940-23 (EudraCT Number)
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Immune Complex-mediated Autoimmune Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- CSL730 (dose 1 with premedication) (Experimental): administered as a single dose by subcutaneous (SC) injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 2 with premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 3 with premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 1 without premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 2 without premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 3 without premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 4 without premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 5 without premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 6 without premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- CSL730 (dose 7 without premedication) (Experimental): administered as a single dose by SC injection or by SC infusion
  Interventions: Biological: CSL730
- Placebo (Placebo Comparator): A solution matching the excipient profile of CSL730 without the active substance administered as a single dose by SC injection or by SC infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSL730 — solution for injection and infusion
  Other Names: Recombinant trivalent human IgG1 Fc multimer
  Arms: CSL730 (dose 1 with premedication); CSL730 (dose 1 without premedication); CSL730 (dose 2 with premedication); CSL730 (dose 2 without premedication); CSL730 (dose 3 with premedication); CSL730 (dose 3 without premedication); CSL730 (dose 4 without premedication); CSL730 (dose 5 without premedication); CSL730 (dose 6 without premedication); CSL730 (dose 7 without premedication)
Drug: Placebo — A solution matching the excipient profile of CSL730 without the active substance
  Arms: Placebo

SUMMARY:
This phase 1, randomized, double-blind, placebo-controlled study will assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending doses of CSL730 administered by subcutaneous (SC) injection or SC infusion in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adult subjects aged ≥ 18 to ≤ 55 years
* Females must be either postmenopausal or sterile
* Body weight between ≥ 50 and ≤ 110 kg and body mass index between ≥ 18.0 kg/m2 and ≤ 30 kg/m2

Exclusion Criteria:

* History or current evidence of a clinically significant medical condition, disorder, or disease, including but not limited to any of the following: hepatic (hepatitis, cirrhosis, or history of liver disease, drug reaction, or aminotransaminase elevations, if known); biliary; renal; cardiac; bronchopulmonary; vascular; hematologic; gastrointestinal; allergy; endocrine / metabolic (diabetes, thyroid disorders, adrenal disease); neurologic (including history of migraine); psychiatric; immunologic; dermatologic; oncologic (subjects with resected cervical or skin cancer [except melanoma] who have had no evidence of disease in the last 5 years are eligible), that precludes designation of healthy subjects as judged by the Investigator
* History or evidence of congenital or acquired immunosuppressive condition(s), including positive serology for human immunodeficiency virus infection or taking immunosuppressive agents.
* Evidence of active or latent tuberculosis
* Hospitalization within 3 months before IP administration or planned hospitalization at any time during the study.
* History of any drug allergy, hypersensitivity (excluding hay fever) or intolerance to latex or any drug product
* A positive test result for drugs of abuse.
* Smokers within 3 months before Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment emergent adverse events (TEAEs) overall, by causality, and by severity | Within 96 hours and up to 56 days after CSL730 administration
Percent of subjects with TEAEs overall, by causality, and by severity | Within 96 hours and up to 56 days after CSL730 administration
Number of subjects with localized administration site AEs overall, by causality, and by severity | Within 96 hours and up to 56 days after CSL730 administration
Percent of subjects with localized administration site AEs overall, by causality, and by severity | Within 96 hours and up to 56 days after CSL730 administration

SECONDARY OUTCOMES:
Maximum concentration (Cmax) for CSL730 in serum samples | up to 56 days after CSL730 administration
Area under the concentration-time curve from time 0 to the last quantifiable time point (AUC0-last) for CSL730 in serum samples | up to 56 days after CSL730 administration
Area under the concentration-time curve from time 0 extrapolated to time infinity (AUC0-inf) for CSL730 in serum samples | up to 56 days after CSL730 administration
Time of maximum concentration (Tmax) for CSL730 in serum samples | up to 56 days after CSL730 administration
Terminal elimination half-life (T1/2) for CSL730 in serum samples | up to 56 days after CSL730 administration
Apparent total systemic clearance (CL/F) for CSL730 in serum samples | up to 56 days after CSL730 administration
Apparent volume of distribution during the elimination phase (Vz/F) for CSL730 in serum samples | up to 56 days after CSL730 administration
Levels of anti-CSL730 antibodies detected in serum samples | Days 15, 29, and 56

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- PAREXEL Early Phase Clinical Unit (London), Northwick Park Hospital, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.